CLINICAL TRIAL: NCT00946647
Title: A Phase Ib/IIb, Open-label, Multi-center, Study of Oral Panobinostat (LBH589) Administered With 5-Azacitidine (in Adult Patients With Myelodysplastic Syndromes (MDS), Chronic Myelomonocytic Leukemia (CMML), or Acute Myeloid Leukemia (AML).
Brief Title: A Phase Ib/IIb, Open-label, Multi-center, Study of Oral Panobinostat Administered With 5-Azacitidine (in Adult Patients With Myelodysplastic Syndromes (MDS), Chronic Myelomonocytic Leukemia (CMML), or Acute Myeloid Leukemia (AML).
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CLBH589H2101; 2009-010548-32 (EudraCT Number)
Record Dates: First submitted 2009-07-07; First posted 2009-07-27 (Estimated); Results first posted 2020-06-23 (Actual); Last update posted 2020-08-04 (Actual); Status verified 2020-07

CONDITIONS: Myelodysplastic Syndromes; Chronic Myelomonocytic Leukemia; Acute Myeloid Leukemia
Keywords: Myelodysplastic Syndromes; Chronic Myelomonocytic Leukemia; Acute Myeloid Leukemia; hypomethylating therapy; deacetylase inhibitor; MDS; CMML; AML
MeSH Terms: conditions — Myelodysplastic Syndromes; Leukemia, Myelomonocytic, Chronic; Leukemia, Myeloid, Acute | interventions — Panobinostat; Azacitidine

STUDY DESIGN:
Masking Description: Treatment was assigned sequentially for the initial dose escalation part (phase Ib): If a dose was safe, the next cohort started with the next dose level. Randomization applies only for the phase IIb part.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes

ARMS (2):
- Panobinostat + 5-Azacytidine (Experimental): In phase I: Panobinostat : Escalating doses starting with 20 mg delivered orally at Day 3, Day 5, Day 8, Day 10, Day 12, Day 15.
  In phase II: Panobinostat : Rapid Phase II doses at 30 mg delivered orally at Day 3, Day 5, Day 8, Day 10, Day 12, Day 15.
  In both phases, dose of 5-Azacytidine was 75 mg/m^2, subcutaneously Daily for Day 1 to Day 7.
  Interventions: Drug: Panobinostat (LBH589); Drug: 5-Azacytidine
- 5-Azacytidine (Active Comparator): The dose of 5-Aza was fixed at 75 mg/m2/day for 7 days in Week 1 of each cycle. 5-Aza was sourced locally, except in 4 countries (Hungary, Switzerland, UK, and Spain, for which a central purchase was used by Novartis.
  Dose of 5-Azacytidine : 75 mg/m^2 subcutaneously daily from Day 1 to Day 7.
  Interventions: Drug: 5-Azacytidine

INTERVENTIONS:
Drug: Panobinostat (LBH589) — Panobinostat was supplied by Novartis as immediate-release hard gelatin capsules in strengths of 5 mg, 10 mg, and 20 mg packaged in high density polyethylene bottles.
  Arms: Panobinostat + 5-Azacytidine
Drug: 5-Azacytidine

SUMMARY:
The purpose of this randomized, two-arm, open-label expansion phase study was to collect preliminary efficacy data of panobinostat at the recommended phase II dose (RPIID) level in combination with azacytidine (5-Aza) versus an active control arm 5-Aza alone. This randomized phase II part also allowed collecting safety data of panobinostat in combination with 5-Aza in comparison to single-agent 5-aza.

DETAILED DESCRIPTION:
The primary objective of the phase lb portion of this study was to determine the maximum tolerated dose (MTD )and/or recommended phase ll dose (RPIID) of oral panobinostat in combination with a fixed dose of 5-Aza in adult patients with International Prognostic Scoring System intermediate-2 (IPSS INT-2) or high risk myelodysplastic syndrome (MDS), Chronic myelomonocytic leukemia (CMML), or Acute myelogenous leukemia (AML).

The primary objective of the phase llb portion of this study was to assess preliminary efficacy of treatment with the panobinostat and 5-Aza combination at the RPIID relative to treatment with single agent 5-Aza through the assessment of composite CR (complete response (CR) or CRi or bone marrow CR).

In the phase lb phase of the study, the patients received escalating oral doses of panobinostat commencing in Cycle 1. The starting dose for panobinostat was 20 mg/day administered orally commencing on Day 3. Each treatment cycle consisted of 28 days (4 weeks). In each cycle, panobinostat was administered twice in Week 1 (Day 3, Day 5), thrice in Week 2 (Day 8, Day 10, and Day 12) and once in Week 3 (Day 15), with no dosing in Week 4. Successive cohorts of patients received escalating doses of panobinostat until the MTD/RPIID was determined. The dose of 5-Aza was fixed at 75 mg/m2/day for 7 days in Week 1 of each cycle.

After the MTD/RPIID was determined, enrollment in the Phase Ib part was closed and the Phase IIb part of the study commenced. Ongoing patients from the Phase Ib part continued their treatment at the assigned dose level according to the regimen and schedule for the Phase Ib part.

Once the RPIID was defined in Phase Ib, additional 80 patients were to be enrolled into the Phase IIb part of the study and randomly assigned in a 1:1 ratio receiving the RPIID of panobinostat plus 5-Aza (investigational arm) or single agent 5-Aza (active control arm). The treatment schedule for the investigational arm was the same as that for the Phase Ib. Single agent 5-Aza (active control arm) was administered according to the locally approved label (75mg/m2 daily for 7 days). Patients continued treatment until disease progression, unacceptable toxicity or consent withdrawal, whichever came first.

ELIGIBILITY:
Inclusion Criteria:

Phase l:

* Patients with cytopathologically confirmed diagnosis of AML according to WHO criteria, excluding acute promyelocytic leukemia who are eligible for Vidaza treatment
* ECOG performance status greater less than or equal to 2

Phase ll:

* Adult patients (age ≥ 18 years) who were candidates for treatment with 5-Aza and present with one of the following:

  * intermediate-2 or high-risk myelodysplastic syndromes according to the International Prognostic Scoring System (IPSS). OR
  * AML with multilineage dysplasia and maximum of 30% blasts (former RAEB-T according to FAB) OR
  * chronic myelomonocytic leukemia (CMML)
* Patients must have had the following laboratory values unless elevations are considered due to MDS or leukemia: AST/SGOT and/or ALT/SGPT ≤ 2.5 x ULN; serum creatinine ≤ 1.5 x ULN; serum bilirubin (total and direct) ≤ 2 x ULN; electrolyte panel within normal ranges (WNL) for the institution.

Exclusion Criteria:

Phase l:

* Prior treatment with deacetylase inhibitors
* Concurrent therapy with any other investigational agent

Phase ll:

* Planned hematopoietic stem-cell transplantation (HSCT)
* Patients with therapy-related MDS
* Patients with therapy-related AML and/or relapsed/refractory AML
* Patients with impaired cardiac function including any of the following:

  * Complete left bundle branch block or use of a permanent cardiac pacemaker, congenital long QT syndrome, history or presence of ventricular tachyarrhythmia, clinically significant resting bradycardia (<50 beats per minute), QTcF > 460 ms on screening ECG, or right bundle branch block + left anterior hemiblock (bifascicular block)
  * Presence of unstable atrial fibrillation (ventricular response rate >100 bpm). Patients with stable atrial fibrillation are eligible provided they do not meet the other cardiac exclusion criteria
  * Previous history of angina pectoris or acute MI within 6 months
  * Screening LVEF <45% by echocardiography or MUGA
  * Other clinically significant heart disease (e.g. uncontrolled hypertension or history of poor compliance with an antihypertensive regimen).
* Any of concurrent severe and/or uncontrolled medical conditions which could compromise participation in the study. For example:

  * Uncontrolled diabetes
  * Active or uncontrolled infection
  * Uncontrolled hypothyroidism
  * Acute or chronic liver or renal disease
* Patient had evidence of clinically significant mucosal or internal bleeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 113 (Actual)
Dates: Start 2009-12-02 (Actual); Primary Completion 2019-04-29 (Actual); Study Completion 2019-04-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (37):
- United States (8):
  - Georgia Health Sciences University Dept. of MCG, Augusta, Georgia
  - Goshen Center for Cancer Care IU Cancer Center, Indianapolis, Indiana
  - University of Kansas Hospital and Medical Center SC - Univ KS, Kansas City, Kansas
  - Dana Farber Cancer Institute Beth Israel Deaconess Med Ctr, Boston, Massachusetts
  - Memorial Sloan Kettering Sloan Kettering 2, New York, New York
  - Cleveland Clinic Foundation Cleve Clinic, Cleveland, Ohio
  - Medical University of South Carolina -Hollings Cancer Center MUSC, Charleston, South Carolina
  - University of Texas MD Anderson Cancer Center Dept of MD Anderson (16), Houston, Texas
- Austria (2):
  - Novartis Investigative Site, Innsbruck
  - Novartis Investigative Site, Vienna
- Belgium (2):
  - Novartis Investigative Site, Bruges
  - Novartis Investigative Site, Yvoir
- Canada (2):
  - Novartis Investigative Site, Edmonton, Alberta
  - Novartis Investigative Site, Toronto, Ontario
- Novartis Investigative Site, Bobigny, France
- Germany (2):
  - Novartis Investigative Site, Frankfurt
  - Novartis Investigative Site, Freiburg im Breisgau
- Hungary (4):
  - Novartis Investigative Site, Budapest
  - Novartis Investigative Site, Debrecen
  - Novartis Investigative Site, Kaposvár
  - Novartis Investigative Site, Szeged
- Italy (3):
  - Novartis Investigative Site, Florence, FI
  - Novartis Investigative Site, Reggio Calabria, RC
  - Novartis Investigative Site, Roma, RM
- South Korea (2):
  - Novartis Investigative Site, Seoul, Korea
  - Novartis Investigative Site, Seoul
- Spain (3):
  - Novartis Investigative Site, Málaga, Andalusia
  - Novartis Investigative Site, Barcelona, Catalonia
  - Novartis Investigative Site, Madrid
- Sweden (2):
  - Novartis Investigative Site, Gothenburg
  - Novartis Investigative Site, Stockholm
- Switzerland (3):
  - Novartis Investigative Site, Basel
  - Novartis Investigative Site, Geneva
  - Novartis Investigative Site, Sankt Gallen
- Novartis Investigative Site, Bangkok, Thailand
- United Kingdom (2):
  - Novartis Investigative Site, London
  - Novartis Investigative Site, Wolverhampton

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent expert panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data is currently available according to the process described on www.clinicalstudydatarequest.com.
URL: https://www.clinicalstudydatarequest.com

REFERENCES:
- [Derived] Garcia-Manero G, Sekeres MA, Egyed M, Breccia M, Graux C, Cavenagh JD, Salman H, Illes A, Fenaux P, DeAngelo DJ, Stauder R, Yee K, Zhu N, Lee JH, Valcarcel D, MacWhannell A, Borbenyi Z, Gazi L, Acharyya S, Ide S, Marker M, Ottmann OG. A phase 1b/2b multicenter study of oral panobinostat plus azacitidine in adults with MDS, CMML or AML with ⩽30% blasts. Leukemia. 2017 Dec;31(12):2799-2806. doi: 10.1038/leu.2017.159. Epub 2017 May 26. PMID 28546581

RESULTS

PARTICIPANT FLOW:
Recruitment Details: In phase l a total of 31 patients were treated with escalating dose of PAN, 20 mg 30 mg & 40 mg. In phase ll a total of 82 patients were actually randomized with 40 patients assigned to PAN+5-Aza and 42 patients assigned to 5-Aza.
Pre-assignment Details: For phase I, approximately 26 patients were planned to be enrolled in cohorts of at least three MTD evaluable patients per dose level.
  For phase ll, approximately 80 patients were planned to be enrolled, 40 patients per arm.
Groups:
- PAN + 5-Aza 20 mg: In this escalating phase, participants took panobinostat of 20 mg delivered orally at Day 3, Day 5, Day 8, Day 10, Day 12, Day 15 and a fixed dose of 5-Azacytidine (5-Aza) at 75 mg/m2/day for 7 days in Week 1 of each cycle.
- PAN + 5-Aza 30 mg: In this escalating phase, participants took panobinostat of 30 mg delivered orally at Day 3, Day 5, Day 8, Day 10, Day 12, Day 15 and a fixed dose of 5-Azacytidine (5-Aza) at 75 mg/m2/day for 7 days in Week 1 of each cycle.
- PAN + 5-Aza 40 mg: In this escalating phase, participants took panobinostat of 40 mg delivered orally at Day 3, Day 5, Day 8, Day 10, Day 12, Day 15 and a fixed dose of 5-Azacytidine (5-Aza) at 75 mg/m2/day for 7 days in Week 1 of each cycle
- Panobinostat + 5-Azacytidine: In phase II: Panobinostat : Rapid Phase II doses at 30 mg delivered orally at Day 3, Day 5, Day 8, Day 10, Day 12, Day 15.
  In both phases, dose of 5-Azacytidine was 75 mg/m^2, subcutaneously Daily for Day 1 to Day 7.
Period: Phase 1 Part
Arm/Group | PAN + 5-Aza 20 mg | PAN + 5-Aza 30 mg | PAN + 5-Aza 40 mg | Panobinostat + 5-Azacytidine | 5-Azacytidine
Started | 6 | 18 | 7 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0
Not Completed | 6 | 18 | 7 | 0 | 0
Not completed — Adverse Event | 2 | 5 | 3 | 0 | 0
Not completed — Disease progression | 3 | 6 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 4 | 3 | 0 | 0
Not completed — Abnormal values | 0 | 2 | 0 | 0 | 0
Not completed — Reason missing | 0 | 1 | 0 | 0 | 0
Period: Phase ll Part
Arm/Group | PAN + 5-Aza 20 mg | PAN + 5-Aza 30 mg | PAN + 5-Aza 40 mg | Panobinostat + 5-Azacytidine | 5-Azacytidine
Started | 0 | 0 | 0 | 40 | 42
Safety Set | 0 | 0 | 0 | 38 (2 pts rand. to this grp did not receive PAN) | 42 (2 pts rand. to PAN+5AZA, did not receive PAN but received 5AZA)
Completed | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 40 | 42
Not completed — Untreated | 0 | 0 | 0 | 0 | 2
Not completed — Adverse Event | 0 | 0 | 0 | 10 | 6
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 8 | 6
Not completed — Administrative problems | 0 | 0 | 0 | 3 | 8
Not completed — Death | 0 | 0 | 0 | 7 | 4
Not completed — Disease progression | 0 | 0 | 0 | 6 | 14
Not completed — Protocol Violation | 0 | 0 | 0 | 4 | 2
Not completed — Subj cond no longer required study drug | 0 | 0 | 0 | 2 | 0

BASELINE CHARACTERISTICS:
Population: Full analysis set: Consisted of all patients who were randomized to one of the two treatment arms
Groups:
- Total: Total of all reporting groups
Arm/Group | PAN + 5-Aza 20 mg | PAN + 5-Aza 30 mg | PAN + 5-Aza 40 mg | Panobinostat + 5-Azacytidine | 5-Azacytidine | Total
Number analyzed (Participants) | 6 | 18 | 7 | 40 | 42 | 113
Age, Customized [Number; unit: participants]
  < 65 | 1 | 5 | 1 | 14 | 8 | 29
  >= 65 | 5 | 13 | 6 | 26 | 34 | 84
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 10 | 4 | 11 | 17 | 44
  Male | 4 | 8 | 3 | 29 | 25 | 69
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 5 | 15 | 6 | 29 | 36 | 91
  Black | 0 | 0 | 1 | 1 | 0 | 2
  Asian | 0 | 0 | 0 | 7 | 2 | 9
  Other | 1 | 3 | 0 | 3 | 4 | 11

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Dose Limiting Toxicity (DLT) (Phase lb)
Description: Dose limiting toxicity (DLT) was defined as a toxicity requiring treatment withdrawal and included the following: Non-hematologic toxicity qualifying for DLT and Hematologic toxicity qualifying for DLT
Time Frame: within the first 28 days (cycle 1)
Population: Maximum Tolerated Dose (MTD) determining set: Consisted of all patients of the safety set who either received sufficient study treatment as defined in the minimum exposure criteria in Cycle 1 (patients had to have 100% of the planned dose of each compound), and had sufficient safety evaluations or discontinued due to DLT in Cycle 1.
Measure: Number; unit: Participants
Arm/Group | PAN + 5-Aza 20 mg | PAN + 5-Aza 30 mg | PAN + 5-Aza 40 mg
Number analyzed (Participants) | 5 | 14 | 7
Participants | 1 | 3 | 2

2. Primary Outcome: Number of Dose Limiting Toxicity (DLT) (Phase lb)
Description: as for outcome 1
Time Frame: within the first 28 days (cycle 1)
Population: as for outcome 1
Measure: Number; unit: DLTs
Arm/Group | PAN + 5-Aza 20 mg | PAN + 5-Aza 30 mg | PAN + 5-Aza 40 mg
Number analyzed (Participants) | 5 | 14 | 7
DLTs | 2 | 6 | 4

3. Primary Outcome: Composite Complete Response (Phase Llb)
Description: Composite complete response is defined as complete response (CR), Complete response with incomplete blood count recovery (CRi) or bone marrow complete response (BM-CR) as defined by the International Working Group (IWG) response criteria.
Time Frame: 48 months
Population: Full analysis set: Consisted of all patients who were randomized to one of the two treatment arms
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Panobinostat + 5-Azacytidine | 5-Azacytidine
Number analyzed (Participants) | 40 | 42
Percentage of participants | 27.5 [14.60 to 43.89] | 14.3 [5.43 to 28.54]

4. Secondary Outcome: Clinical Response Other Than Composite Clinical Response for Myeloid Dysplastic Syndromes(MDS)/Chronic Myelomonocytic Leukemia (CMML) Patients Per Investigator (Phase Llb)
Description: This is the best overall response as measured by Clinical response. Clinical response is defined as having complete remission (CR), bone marrow complete remission (BM-CR), partial remission or hematologic improvement (HI) as defined by the International Working Group (IWG) response criteria.
Time Frame: 48 months
Population: Full analysis set: Consisted of all patients who were randomized to one of the two treatment arms
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Panobinostat + 5-Azacytidine | 5-Azacytidine
Number analyzed (Participants) | 31 | 29
Percentage of participants | 41.9 [24.5 to 60.9] | 41.4 [23.5 to 61.1]

5. Secondary Outcome: Clinical Response Other Than Composite Clinical Response for Acute Myelogenous Leukemia (AML) Patients Per Investigator (Phase Llb)
Description: This is the best overall response as measured by Clinical response. Clinical response is defined as having complete remission (CR), complete remission with incomplete blood count recovery (CRi) or partial remission as defined by the International Working Group (IWG) response criteria.
Time Frame: 48 months
Population: Full analysis set: Consisted of all patients who were randomized to one of the two treatment arms
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Panobinostat + 5-Azacytidine | 5-Azacytidine
Number analyzed (Participants) | 9 | 13
Percentage of participants | 22.2 [2.8 to 60.0] | 30.8 [9.1 to 61.4]

6. Secondary Outcome: Overall Response Rate (ORR) Assessed by Best Overall Response: Participants With MDS/CMML Per Investigator (Phase Llb)
Description: Best overall response as measured by complete remission (CR) or bone marrow CR (BM-CR) or partial remission (PR) or hematologic improvement (HI).
  Overall response patients achieved other than the composite CR by individual response category: CR, CRi, mCR or PR as defined by the International Working Group (IWG) response criteria.
Time Frame: 48 months
Population: Full analysis set (FAS): Consisted of all patients who were randomized to one of the two treatment arms.
Measure: Number; unit: Percentage of participants
Arm/Group | Panobinostat + 5-Azacytidine | 5-Azacytidine
Number analyzed (Participants) | 31 | 29
Percentage of participants
  Clinical response (CR, BM-CR, PR, HI) | 41.9 | 41.4
  Complete remission (CR) | 16.1 | 6.9
  Bone marrow CR (BM-CR) | 12.9 | 3.4
  Partial remission (PR) | 0.0 | 6.9

7. Secondary Outcome: Overall Response Rate (ORR) Assessed by Best Overall Response: Participants With AML Per Investigator (Phase Llb)
Description: Best overall response as measured by complete remission (CR) or complete response with incomplete blood count recovery (CRi) or partial remission (PR).
  Overall response patients achieved other than the composite CR by individual response category: CR, CRi or PR.
Time Frame: 48 months
Population: Full analysis set (FAS): Consisted of all patients who were randomized to one of the two treatment arms.
Measure: Number; unit: Percentage of participants
Arm/Group | Panobinostat + 5-Azacytidine | 5-Azacytidine
Number analyzed (Participants) | 9 | 13
Percentage of participants
  Clinical response (CR, CRi, PR) | 22.2 | 30.8
  Complete remission (CR) | 11.1 | 15.4
  Compl remiss. with incompl blood cnt recovery(CRi) | 11.1 | 7.7
  Partial remission (PR) | 0.0 | 7.7

8. Secondary Outcome: Hematologic Improvement (HI) for Myeloid Dysplastic Syndromes(MDS)/Chronic Myelomonocytic Leukemia (CMML) Patients Per Investigator (Phase Llb)
Description: Hematologic response consists of Erythroid response (HI-E), Platelet response (HI-P) and Neutrophil response (HI-N).
  HI-E: Hgb increase by ≥ 1.5 g/dL over pretreatment & relevant reduction of units of RBC transfusions by an absolute number of at least 4 units of PRBCs/8 weeks compared with the pretreatment transfusion number in the previous 8 weeks. Only RBC transfusions given for a Hgb of ≤ 9.0 g/dL pretreatment will count in the RBC transfusion response evaluation.
  HI-P: Absolute increase of ≥ 30 x 109/L over pretreatment or patients starting with ≥ 20 x 109/L platelets OR increase from <20 x 109/L at pretreatment to > 20 x 109/L and by at least 100%.
  HI-N: At least 100% increase and an absolute increase > 0.5 x 109/L over pretreatment value.
Time Frame: 48 months
Population: Full analysis set: Consisted of all patients who were randomized to one of the two treatment arms
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Panobinostat + 5-Azacytidine | 5-Azacytidine
Number analyzed (Participants) | 31 | 29
Percentage of participants
  Erythroid response (HI-E) | 25.8 [11.9 to 44.6] | 31.0 [15.3 to 50.8]
  Platelet response (HI-P) | 35.5 [19.2 to 54.6] | 24.1 [10.3 to 43.5]
  Neutrophil response (HI-N) | 19.4 [7.5 to 37.5] | 13.8 [3.9 to 31.7]

9. Secondary Outcome: 1-year Survival Rate (Phase Llb)
Description: Overall survival was defined as the time from date of randomization to date of death due to any cause. If a patient was not known to have died, survival was censored at the date of last contact. Patients not known to have died were censored for 'Lost to follow-up' if the time between their last contact date and the analysis cut-off date was longer than 3 months and 2 weeks (104 days) during the first year after study evaluation completion, and longer than 6 months and 2 weeks (194 days), thereafter. The 1-year survival rate was obtained from the Kaplan-Meier analysis of overall survival, and its variance was estimated by Greenwood's formula.
Time Frame: 12 months
Population: Full analysis set: Consisted of all patients who were randomized to one of the two treatment arms
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Panobinostat + 5-Azacytidine | 5-Azacytidine
Number analyzed (Participants) | 40 | 42
months | 14.9 [10.4 to NA] — NA - The follow-up was too short that the quantiles of the survival distribution could not be estimated. | 15.6 [11.4 to NA] — NA - The follow-up was too short that the quantiles of the survival distribution could not be estimated.

10. Secondary Outcome: Time to Progression (TTP) (Phase Llb)
Description: Time to progression (TTP) was defined as the time from the date of randomization to the date of the first documented PD per investigator's assessment or death due to study indication.
  Time to progression was analyzed by the Kaplan Meier method. Based on the Guidelines for Implementation of international working group (IWG) response criteria in AML, MDS and CMML according to Cheson 2003 and 2006.
Time Frame: 48 months
Population: Full analysis set: Consisted of all patients who were randomized to one of the two treatment arms
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Panobinostat + 5-Azacytidine | 5-Azacytidine
Number analyzed (Participants) | 40 | 42
months | NA [11.1 to NA] — NA - The follow-up was too short that the quantiles of the survival distribution could not be estimated. | 15.2 [11.0 to NA] — NA - The follow-up was too short that the quantiles of the survival distribution could not be estimated.

ADVERSE EVENTS:
Time Frame: Adverse Event (AE) timeframe: Adverse events were collected from first dose of study treatment until end of study treatment plus 28 days post treatment, up to maximum duration 397.1 weeks.
Description: Adverse Event (AE): Any sign or symptom that occurs during the study treatment plus the 28 days post treatment.
  2 patients randomized to PAN+5AZA received only 5AZA & no PAN & were part of the safety set for 5AZA group. Also, 2 patients rand. to 5AZA did not receive any treatment & were not part of the safety set but were part of the FAS for the 5AZA group
Groups:
- Phase Ib PAN + 5-Aza 20mg: In this escalating phase, participants took panobinostat of 20 mg delivered orally at Day 3, Day 5, Day 8, Day 10, Day 12, Day 15 and a fixed dose of 5-Azacytidine (5-Aza) at 75 g/m2/day for 7 days in Week 1 of each cycle
- Phase Ib PAN + 5-Aza 30mg: In this escalating phase, participants took panobinostat of 30 mg delivered orally at Day 3, Day 5, Day 8, Day 10, Day 12, Day 15 and a fixed dose of 5-Azacytidine (5-Aza) at 75 mg/m2/day for 7 days in Week 1 of each cycle
- Phase Ib PAN + 5-Aza 40mg: In this escalating phase, participants took panobinostat of 40 mg delivered orally at Day 3, Day 5, Day 8, Day 10, Day 12, Day 15 and a fixed dose of 5-Azacytidine (5-Aza) at 75 mg/m2/day for 7 days in Week 1 of each cycle
- Phase IIb PAN + 5-Aza: In phase II: Panobinostat : Rapid Phase II doses at 30 mg delivered orally at Day 3, Day 5, Day 8, Day 10, Day 12, Day 15.
  In both phases, dose of 5-Azacytidine was 75 mg/m^2, subcutaneously Daily for Day 1 to Day 7.
- Phase IIb 5-Aza: The dose of 5-Aza was fixed at 75 mg/m2/day for 7 days in Week 1 of each cycle. 5-Aza was sourced locally, except in 4 countries (Hungary, Switzerland, UK, and Spain, for which a central purchase was used by Novartis.
  Dose of 5-Azacytidine: 75 mg/m^2 subcutaneously daily from Day 1 to Day
- Phase Ib and IIb: Patients in the Panobinostat + 5-Azacytidine arm and in the 5-Azacytidine arm
Arm/Group | Phase Ib PAN + 5-Aza 20mg | Phase Ib PAN + 5-Aza 30mg | Phase Ib PAN + 5-Aza 40mg | Phase IIb PAN + 5-Aza | Phase IIb 5-Aza | Phase Ib and IIb
All-Cause Mortality (participants affected / at risk) | 0/6 | 1/18 | 2/7 | 6/38 | 3/42 | 12/111
Serious Adverse Events (participants affected / at risk) | 5/6 | 15/18 | 6/7 | 28/38 | 28/42 | 82/111
Other Adverse Events (participants affected / at risk) | 6/6 | 18/18 | 7/7 | 38/38 | 38/42 | 107/111
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase Ib PAN + 5-Aza 20mg (N=6) | Phase Ib PAN + 5-Aza 30mg (N=18) | Phase Ib PAN + 5-Aza 40mg (N=7) | Phase IIb PAN + 5-Aza (N=38) | Phase IIb 5-Aza (N=42) | Phase Ib and IIb (N=111)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 2 | 0 | 2
Anaemia of malignant disease (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 2 | 6 | 3 | 10 | 6 | 27
Haemolytic anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 1
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 2 | 2 | 5
Pancytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 1 | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 3 | 3 | 7
Acute myocardial infarction (Cardiac disorders) | 0 | 1 | 0 | 1 | 0 | 2
Angina pectoris (Cardiac disorders) | 0 | 1 | 0 | 0 | 1 | 2
Atrial fibrillation (Cardiac disorders) | 1 | 1 | 1 | 0 | 0 | 3
Atrial flutter (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 1
Cardiac failure (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 1
Cardio-respiratory arrest (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 1
Coronary artery disease (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 1
Left ventricular hypertrophy (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 1
Myocarditis (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 1
Diplopia (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 1
Uveitis (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 1
Vision blurred (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 1
Colitis (Gastrointestinal disorders) | 0 | 2 | 0 | 1 | 0 | 3
Constipation (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 0 | 2
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 1 | 3
Duodenitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 1
Gastritis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 1
Gastroenteritis eosinophilic (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 1 | 3
Large intestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 1
Melaena (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 2 | 2
Nausea (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 0 | 2
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 1
Tongue haematoma (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 1
Volvulus (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 0 | 2
Asthenia (General disorders) | 2 | 0 | 2 | 0 | 0 | 4
Death (General disorders) | 0 | 0 | 0 | 1 | 0 | 1
Fatigue (General disorders) | 0 | 1 | 0 | 0 | 0 | 1
Pyrexia (General disorders) | 0 | 2 | 0 | 3 | 0 | 5
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0 | 1
Abscess soft tissue (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1
Bacteraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1
Bacterial sepsis (Infections and infestations) | 0 | 1 | 0 | 1 | 0 | 2
Breast cellulitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 1
Bronchopulmonary aspergillosis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1
Cellulitis (Infections and infestations) | 0 | 1 | 0 | 1 | 2 | 4
Diverticulitis (Infections and infestations) | 0 | 1 | 0 | 0 | 1 | 2
Erysipelas (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 1
Escherichia bacteraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1
Escherichia infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 1
Gastrointestinal infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 1
Herpes simplex (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1
Impetigo (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 1
Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1
Lower respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1
Lung infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 1
Neutropenic sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 3 | 3
Oral bacterial infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 1
Parotitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1
Perirectal abscess (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 1
Pharyngeal abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1
Pneumonia (Infections and infestations) | 0 | 2 | 2 | 8 | 4 | 16
Pulmonary sepsis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 1
Sepsis (Infections and infestations) | 0 | 1 | 0 | 4 | 4 | 9
Septic shock (Infections and infestations) | 1 | 0 | 1 | 2 | 0 | 4
Sinusitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 1
Staphylococcal sepsis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 1
Tooth infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1
Urinary tract infection (Infections and infestations) | 0 | 1 | 0 | 1 | 0 | 2
Femur fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 1
Hip fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 1
Skin laceration (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 1
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 1
Transfusion reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 1
Ulna fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 1
Blood creatine phosphokinase increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 1
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 1
Electrocardiogram ST segment depression (Investigations) | 0 | 0 | 0 | 1 | 0 | 1
Electrocardiogram T wave inversion (Investigations) | 0 | 1 | 0 | 1 | 0 | 2
Gamma-glutamyltransferase increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 1
Haemoglobin decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 1
Heart rate increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 1
Troponin T increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 2 | 0 | 0 | 1 | 3
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 1 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 1 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 0 | 0 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 1
Benign anorectal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 1
Large cell lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 1
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 1
Cerebral haemorrhage (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 1
Dysarthria (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 1
Haemorrhage intracranial (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 1
Headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 2 | 2
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 1 | 1 | 0 | 0 | 2
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 1
Prerenal failure (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 1
Renal failure (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 1
Urinary retention (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 2 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 1 | 2
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 0 | 2
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 1 | 2
Angioedema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 1
Embolism venous (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 1
Haematoma (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 1
Hypotension (Vascular disorders) | 0 | 1 | 0 | 0 | 1 | 2
Peripheral artery occlusion (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Phase Ib PAN + 5-Aza 20mg (N=6) | Phase Ib PAN + 5-Aza 30mg (N=18) | Phase Ib PAN + 5-Aza 40mg (N=7) | Phase IIb PAN + 5-Aza (N=38) | Phase IIb 5-Aza (N=42) | Phase Ib and IIb (N=111)
Anaemia (Blood and lymphatic system disorders) | 2 | 8 | 4 | 12 | 14 | 40
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 3 | 0 | 6 | 2 | 11
Leukocytosis (Blood and lymphatic system disorders) | 0 | 2 | 0 | 0 | 1 | 3
Leukopenia (Blood and lymphatic system disorders) | 1 | 4 | 1 | 4 | 1 | 11
Lymphopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 2 | 0 | 2
Neutropenia (Blood and lymphatic system disorders) | 2 | 8 | 3 | 16 | 10 | 39
Pancytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 3 | 1 | 4
Splenomegaly (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 3 | 12 | 4 | 18 | 10 | 47
Thrombocytosis (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 2 | 3
Thrombotic microangiopathy (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 1
Angina pectoris (Cardiac disorders) | 1 | 1 | 0 | 1 | 0 | 3
Arrhythmia (Cardiac disorders) | 1 | 0 | 0 | 0 | 1 | 2
Atrial fibrillation (Cardiac disorders) | 1 | 1 | 2 | 3 | 1 | 8
Atrial flutter (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 1
Bundle branch block left (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 1
Cardiac failure acute (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 1
Extrasystoles (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 1
Hypertensive heart disease (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 1
Myocarditis (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 1
Palpitations (Cardiac disorders) | 0 | 3 | 0 | 0 | 0 | 3
Pericardial effusion (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 1
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 1 | 2 | 0 | 3
Tachycardia (Cardiac disorders) | 1 | 1 | 2 | 0 | 1 | 5
Ventricular extrasystoles (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 1
Ear disorder (Ear and labyrinth disorders) | 0 | 0 | 1 | 0 | 0 | 1
Ear pain (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 2 | 3
Hypoacusis (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 1 | 2
Otorrhoea (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 0 | 1
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 1 | 0 | 0 | 1
Vertigo (Ear and labyrinth disorders) | 1 | 2 | 0 | 0 | 1 | 4
Hypothyroidism (Endocrine disorders) | 1 | 0 | 0 | 0 | 0 | 1
Thyroid disorder (Endocrine disorders) | 0 | 1 | 0 | 0 | 0 | 1
Blepharitis (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 1
Cataract (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 1
Diplopia (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 1
Eye irritation (Eye disorders) | 0 | 2 | 0 | 0 | 0 | 2
Optic atrophy (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 1
Pupillary reflex impaired (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 1
Vision blurred (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 1
Visual impairment (Eye disorders) | 1 | 0 | 0 | 1 | 0 | 2
Abdominal distension (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 3 | 6 | 1 | 6 | 2 | 18
Abdominal pain upper (Gastrointestinal disorders) | 1 | 4 | 1 | 2 | 2 | 10
Abdominal wall haematoma (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0 | 2
Abdominal wall mass (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 1
Anal fistula (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 1
Anal incontinence (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0 | 2
Anal skin tags (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0 | 2
Angina bullosa haemorrhagica (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 1 | 3
Ascites (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 2 | 11 | 3 | 10 | 16 | 42
Diarrhoea (Gastrointestinal disorders) | 4 | 15 | 4 | 22 | 9 | 54
Dry mouth (Gastrointestinal disorders) | 0 | 1 | 1 | 3 | 0 | 5
Dyschezia (Gastrointestinal disorders) | 1 | 2 | 0 | 0 | 0 | 3
Dyspepsia (Gastrointestinal disorders) | 1 | 2 | 1 | 0 | 1 | 5
Dysphagia (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0 | 2
Epigastric discomfort (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0 | 2
Flatulence (Gastrointestinal disorders) | 1 | 3 | 0 | 0 | 2 | 6
Gastritis (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 0 | 2
Gastroenteritis eosinophilic (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 1
Gastrointestinal oedema (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 1
Gastrointestinal pain (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 1 | 2 | 1 | 4
Gingival bleeding (Gastrointestinal disorders) | 1 | 3 | 0 | 1 | 1 | 6
Gingival pain (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1 | 2
Haematochezia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 1
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0 | 2
Haemorrhoids (Gastrointestinal disorders) | 2 | 2 | 1 | 5 | 1 | 11
Intra-abdominal haematoma (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 1
Lip swelling (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 1
Loose tooth (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1 | 2
Melaena (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 1
Mouth haemorrhage (Gastrointestinal disorders) | 0 | 3 | 0 | 1 | 2 | 6
Mouth ulceration (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 1 | 3
Nausea (Gastrointestinal disorders) | 4 | 14 | 7 | 23 | 18 | 66
Noninfective gingivitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 1
Parotid gland enlargement (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1 | 2
Proctalgia (Gastrointestinal disorders) | 1 | 2 | 0 | 0 | 0 | 3
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 1 | 1 | 0 | 3
Retroperitoneal haematoma (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 1
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 4 | 6
Swollen tongue (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 1
Tongue coated (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 1
Tooth impacted (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 1
Toothache (Gastrointestinal disorders) | 0 | 3 | 1 | 1 | 3 | 8
Vomiting (Gastrointestinal disorders) | 5 | 9 | 4 | 16 | 12 | 46
Asthenia (General disorders) | 2 | 6 | 1 | 10 | 6 | 25
Catheter site discharge (General disorders) | 0 | 1 | 0 | 0 | 0 | 1
Catheter site erythema (General disorders) | 0 | 0 | 1 | 0 | 0 | 1
Catheter site haematoma (General disorders) | 0 | 1 | 0 | 0 | 0 | 1
Catheter site pain (General disorders) | 0 | 1 | 0 | 0 | 0 | 1
Catheter site phlebitis (General disorders) | 0 | 1 | 0 | 0 | 0 | 1
Chest pain (General disorders) | 0 | 2 | 0 | 0 | 0 | 2
Chills (General disorders) | 0 | 4 | 2 | 3 | 3 | 12
Extravasation (General disorders) | 0 | 0 | 1 | 0 | 0 | 1
Facial pain (General disorders) | 0 | 1 | 1 | 0 | 0 | 2
Fatigue (General disorders) | 4 | 12 | 6 | 10 | 16 | 48
Feeling cold (General disorders) | 1 | 0 | 0 | 0 | 0 | 1
Feeling hot (General disorders) | 0 | 0 | 1 | 0 | 0 | 1
Gait disturbance (General disorders) | 0 | 1 | 2 | 0 | 0 | 3
General physical health deterioration (General disorders) | 0 | 2 | 0 | 1 | 0 | 3
Generalised oedema (General disorders) | 1 | 1 | 0 | 1 | 0 | 3
Injection site bruising (General disorders) | 0 | 1 | 0 | 1 | 0 | 2
Injection site erythema (General disorders) | 0 | 5 | 0 | 3 | 3 | 11
Injection site haematoma (General disorders) | 0 | 1 | 0 | 0 | 0 | 1
Injection site haemorrhage (General disorders) | 0 | 2 | 0 | 1 | 0 | 3
Injection site irritation (General disorders) | 0 | 1 | 0 | 0 | 0 | 1
Injection site pain (General disorders) | 1 | 5 | 0 | 2 | 3 | 11
Injection site pruritus (General disorders) | 0 | 0 | 1 | 0 | 0 | 1
Injection site rash (General disorders) | 1 | 1 | 0 | 2 | 1 | 5
Injection site reaction (General disorders) | 0 | 2 | 1 | 3 | 2 | 8
Localised oedema (General disorders) | 0 | 1 | 0 | 0 | 0 | 1
Malaise (General disorders) | 1 | 0 | 0 | 1 | 4 | 6
Mass (General disorders) | 0 | 0 | 1 | 0 | 0 | 1
Mucosal inflammation (General disorders) | 1 | 0 | 0 | 0 | 0 | 1
Non-cardiac chest pain (General disorders) | 2 | 2 | 1 | 4 | 2 | 11
Oedema peripheral (General disorders) | 2 | 4 | 4 | 8 | 9 | 27
Pain (General disorders) | 1 | 0 | 2 | 2 | 1 | 6
Peripheral swelling (General disorders) | 0 | 2 | 1 | 1 | 1 | 5
Puncture site erythema (General disorders) | 1 | 0 | 0 | 0 | 2 | 3
Pyrexia (General disorders) | 2 | 8 | 4 | 18 | 9 | 41
Swelling (General disorders) | 0 | 1 | 0 | 0 | 0 | 1
Thirst (General disorders) | 0 | 0 | 1 | 1 | 0 | 2
Hepatomegaly (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0 | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0 | 1
Allergic oedema (Immune system disorders) | 0 | 1 | 0 | 0 | 0 | 1
Allergy to chemicals (Immune system disorders) | 0 | 1 | 0 | 0 | 0 | 1
Drug hypersensitivity (Immune system disorders) | 0 | 2 | 0 | 2 | 0 | 4
Hypersensitivity (Immune system disorders) | 0 | 1 | 0 | 0 | 0 | 1
Anal abscess (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 1
Anal fungal infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 1
Anal infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 1
Bacterial infection (Infections and infestations) | 1 | 0 | 1 | 0 | 0 | 2
Bronchitis (Infections and infestations) | 0 | 1 | 0 | 2 | 2 | 5
Candida infection (Infections and infestations) | 1 | 1 | 3 | 0 | 1 | 6
Carbuncle (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 1
Cellulitis (Infections and infestations) | 0 | 2 | 0 | 1 | 4 | 7
Chronic sinusitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 1
Clostridium difficile colitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 1
Clostridium difficile infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 1
Conjunctivitis (Infections and infestations) | 0 | 1 | 0 | 3 | 0 | 4
Device related infection (Infections and infestations) | 0 | 1 | 0 | 0 | 1 | 2
Diverticulitis (Infections and infestations) | 0 | 2 | 0 | 0 | 0 | 2
Enterobacter infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 1
Enterococcal infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 1
Folliculitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 1
Fungal infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 1
Fungal skin infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 1
Haemorrhoid infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 1
Herpes simplex (Infections and infestations) | 0 | 0 | 0 | 2 | 2 | 4
Herpes zoster (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 1
Human polyomavirus infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 1
Infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 1
Infectious colitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 1
Influenza (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 1
Localised infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 1
Mucormycosis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 1
Nasopharyngitis (Infections and infestations) | 0 | 1 | 0 | 1 | 1 | 3
Oral candidiasis (Infections and infestations) | 0 | 1 | 0 | 1 | 2 | 4
Oral herpes (Infections and infestations) | 1 | 3 | 0 | 1 | 2 | 7
Pneumonia (Infections and infestations) | 0 | 2 | 0 | 1 | 3 | 6
Pseudomonas infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 1
Puncture site infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 1
Respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 1
Rhinitis (Infections and infestations) | 0 | 1 | 1 | 2 | 0 | 4
Sinusitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 1
Skin infection (Infections and infestations) | 0 | 3 | 0 | 2 | 1 | 6
Staphylococcal infection (Infections and infestations) | 1 | 1 | 1 | 1 | 1 | 5
Tooth abscess (Infections and infestations) | 0 | 0 | 1 | 1 | 0 | 2
Tooth infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 3 | 3 | 7
Urinary tract infection (Infections and infestations) | 0 | 2 | 1 | 3 | 4 | 10
Wound infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 1
Allergic transfusion reaction (Injury, poisoning and procedural complications) | 0 | 3 | 1 | 1 | 0 | 5
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 3 | 0 | 0 | 0 | 3
Contusion (Injury, poisoning and procedural complications) | 0 | 2 | 2 | 3 | 2 | 9
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 2 | 0 | 0 | 2
Post procedural haematoma (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 1
Post procedural swelling (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 1
Procedural hypertension (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 1
Procedural pain (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 0 | 2 | 4
Tongue injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 1
Tooth fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 1
Transfusion reaction (Injury, poisoning and procedural complications) | 0 | 2 | 3 | 0 | 1 | 6
Activated partial thromboplastin time prolonged (Investigations) | 0 | 0 | 1 | 1 | 0 | 2
Alanine aminotransferase increased (Investigations) | 0 | 2 | 1 | 3 | 2 | 8
Aspartate aminotransferase increased (Investigations) | 0 | 2 | 1 | 4 | 1 | 8
Blood albumin decreased (Investigations) | 0 | 0 | 0 | 2 | 1 | 3
Blood bicarbonate decreased (Investigations) | 0 | 0 | 1 | 0 | 0 | 1
Blood bilirubin increased (Investigations) | 0 | 2 | 0 | 0 | 0 | 2
Blood creatinine decreased (Investigations) | 0 | 0 | 1 | 0 | 0 | 1
Blood creatinine increased (Investigations) | 1 | 5 | 4 | 4 | 0 | 14
Blood folate decreased (Investigations) | 0 | 0 | 1 | 0 | 0 | 1
Blood magnesium decreased (Investigations) | 0 | 0 | 1 | 0 | 0 | 1
Blood phosphorus decreased (Investigations) | 0 | 0 | 1 | 0 | 0 | 1
Blood potassium increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 1
Blood thyroid stimulating hormone decreased (Investigations) | 1 | 0 | 0 | 0 | 0 | 1
Blood urine present (Investigations) | 1 | 1 | 0 | 0 | 0 | 2
Breath sounds abnormal (Investigations) | 0 | 1 | 0 | 1 | 0 | 2
C-reactive protein increased (Investigations) | 1 | 2 | 2 | 2 | 1 | 8
Coagulation test abnormal (Investigations) | 1 | 0 | 0 | 0 | 0 | 1
Electrocardiogram QT prolonged (Investigations) | 0 | 1 | 1 | 3 | 0 | 5
Electrocardiogram T wave abnormal (Investigations) | 0 | 1 | 0 | 0 | 0 | 1
Fibrin D dimer increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 1
Glucose urine present (Investigations) | 0 | 0 | 1 | 0 | 0 | 1
Haemoglobin decreased (Investigations) | 0 | 0 | 0 | 2 | 1 | 3
Left ventricular end-diastolic pressure increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 1
Neutrophil count decreased (Investigations) | 0 | 1 | 1 | 6 | 3 | 11
Nitrite urine present (Investigations) | 0 | 0 | 1 | 0 | 0 | 1
Platelet count decreased (Investigations) | 0 | 1 | 0 | 8 | 2 | 11
Protein urine present (Investigations) | 0 | 0 | 1 | 0 | 0 | 1
Prothrombin time prolonged (Investigations) | 0 | 0 | 1 | 1 | 0 | 2
Prothrombin time shortened (Investigations) | 0 | 0 | 1 | 0 | 0 | 1
Troponin I increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 1
Troponin T increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 1
Urine output decreased (Investigations) | 0 | 0 | 2 | 0 | 0 | 2
Urobilinogen urine increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 1
Vitamin D decreased (Investigations) | 2 | 0 | 0 | 0 | 0 | 2
Weight decreased (Investigations) | 1 | 1 | 1 | 7 | 6 | 16
White blood cell count decreased (Investigations) | 0 | 0 | 0 | 4 | 0 | 4
White blood cells urine positive (Investigations) | 0 | 0 | 1 | 0 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 3 | 6 | 5 | 9 | 6 | 29
Dehydration (Metabolism and nutrition disorders) | 0 | 3 | 3 | 3 | 1 | 10
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 1
Fluid overload (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 3 | 3
Fluid retention (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 1
Gout (Metabolism and nutrition disorders) | 0 | 1 | 1 | 0 | 0 | 2
Hypercreatininaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 2 | 3 | 2 | 0 | 7
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 2 | 1 | 1 | 3 | 7
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 1 | 2
Hypermagnesaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 1
Hyperuricaemia (Metabolism and nutrition disorders) | 1 | 5 | 1 | 2 | 1 | 10
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 1 | 2 | 0 | 1 | 4
Hypocalcaemia (Metabolism and nutrition disorders) | 3 | 7 | 2 | 2 | 2 | 16
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 10 | 3 | 7 | 6 | 27
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 3 | 2 | 2 | 2 | 10
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1 | 3 | 2 | 1 | 7
Hypophosphataemia (Metabolism and nutrition disorders) | 1 | 1 | 2 | 4 | 1 | 9
Iron overload (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 5 | 1 | 3 | 4 | 14
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 2 | 2 | 5 | 4 | 14
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 2 | 2 | 0 | 0 | 5
Coccydynia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 1
Joint effusion (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 1
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1 | 0 | 2
Limb discomfort (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 1
Muscle fatigue (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1 | 1 | 3
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 2 | 1 | 1 | 2 | 6
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1 | 0 | 1 | 4
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 3 | 1 | 2 | 3 | 10
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 3 | 2 | 5
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0 | 1 | 3
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 4 | 2 | 4 | 2 | 13
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 1
Spinal deformity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 1
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 1 | 2
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 1 | 2
Temporomandibular joint syndrome (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 1
Benign lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 1
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 1
Balance disorder (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 1
Disturbance in attention (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 1 | 4 | 2 | 5 | 3 | 15
Dysgeusia (Nervous system disorders) | 2 | 4 | 1 | 3 | 2 | 12
Dyskinesia (Nervous system disorders) | 0 | 0 | 1 | 1 | 0 | 2
Facial paresis (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 1
Headache (Nervous system disorders) | 2 | 4 | 4 | 7 | 7 | 24
Hypotonia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 1
Neuralgia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 1
Normal pressure hydrocephalus (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 1
Paraesthesia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 1
Partial seizures (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 1
Polyneuropathy (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 1
Sciatica (Nervous system disorders) | 1 | 0 | 0 | 0 | 1 | 2
Somnolence (Nervous system disorders) | 1 | 0 | 2 | 0 | 0 | 3
Subarachnoid haemorrhage (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 1
Syncope (Nervous system disorders) | 0 | 2 | 0 | 2 | 2 | 6
Tremor (Nervous system disorders) | 0 | 1 | 0 | 0 | 1 | 2
Agitation (Psychiatric disorders) | 1 | 0 | 0 | 1 | 0 | 2
Anxiety (Psychiatric disorders) | 0 | 1 | 2 | 1 | 1 | 5
Confusional state (Psychiatric disorders) | 0 | 1 | 2 | 1 | 0 | 4
Delirium (Psychiatric disorders) | 0 | 0 | 0 | 2 | 0 | 2
Depression (Psychiatric disorders) | 0 | 2 | 0 | 1 | 0 | 3
Disorientation (Psychiatric disorders) | 1 | 0 | 1 | 0 | 0 | 2
Fear (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 1
Insomnia (Psychiatric disorders) | 1 | 3 | 3 | 5 | 3 | 15
Personality change (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 1
Sleep disorder (Psychiatric disorders) | 1 | 0 | 0 | 0 | 1 | 2
Anuria (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 1
Bladder pain (Renal and urinary disorders) | 1 | 1 | 0 | 0 | 0 | 2
Dysuria (Renal and urinary disorders) | 0 | 1 | 0 | 2 | 0 | 3
Haematuria (Renal and urinary disorders) | 0 | 0 | 2 | 0 | 0 | 2
Haemorrhage urinary tract (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 1
Renal failure (Renal and urinary disorders) | 0 | 0 | 1 | 1 | 0 | 2
Renal pain (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 1
Urinary incontinence (Renal and urinary disorders) | 1 | 0 | 1 | 0 | 0 | 2
Urinary retention (Renal and urinary disorders) | 0 | 1 | 1 | 0 | 0 | 2
Scrotal erythema (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 1
Scrotal oedema (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 1
Scrotal pain (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 1
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 1 | 1 | 0 | 0 | 2
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 1
Bronchial disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 1
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 1 | 2
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 1
Bronchostenosis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 6 | 2 | 7 | 6 | 23
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 0 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 6 | 3 | 2 | 4 | 18
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 1 | 1 | 4
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 4 | 2 | 5 | 6 | 19
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 1 | 2
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 0 | 2
Hyperventilation (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0 | 0 | 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 2 | 4
Laryngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 1
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 1 | 0 | 0 | 3
Oropharyngeal blistering (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 | 3 | 3 | 0 | 5 | 14
Pharyngeal erythema (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 2 | 1 | 1 | 7
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0 | 3 | 5
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0 | 0 | 2
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1 | 0 | 0 | 3
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2 | 1 | 3
Rhonchi (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 0 | 2
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0 | 1 | 3
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 1
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 2 | 2 | 0 | 0 | 5
Angioedema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 1
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 | 1 | 1 | 0 | 0 | 3
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1 | 0 | 2
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 2 | 1 | 1 | 0 | 2 | 6
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 2 | 0 | 2
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 2 | 1 | 5
Eczema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1 | 0 | 2
Erythema (Skin and subcutaneous tissue disorders) | 1 | 3 | 1 | 1 | 4 | 10
Exfoliative rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1 | 0 | 2
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 2 | 0 | 0 | 0 | 3
Koebner phenomenon (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 1
Nail disorder (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 1
Night sweats (Skin and subcutaneous tissue disorders) | 1 | 2 | 1 | 0 | 0 | 4
Pain of skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 2 | 0 | 2
Papule (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 1
Petechiae (Skin and subcutaneous tissue disorders) | 0 | 7 | 2 | 3 | 1 | 13
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 4 | 3 | 9
Psoriasis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 1
Purpura (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 0 | 1 | 3
Rash (Skin and subcutaneous tissue disorders) | 0 | 4 | 2 | 6 | 4 | 16
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 1 | 2
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 2 | 1 | 5
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1 | 1 | 3
Skin haemorrhage (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 1 | 2
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 1 | 0 | 3
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 1
Skin plaque (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0 | 0 | 2
Swelling face (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 4 | 0 | 5
Arteriosclerosis (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 1
Flushing (Vascular disorders) | 0 | 1 | 0 | 1 | 0 | 2
Haematoma (Vascular disorders) | 0 | 3 | 1 | 2 | 5 | 11
Hypertension (Vascular disorders) | 0 | 4 | 0 | 0 | 1 | 5
Hypotension (Vascular disorders) | 2 | 2 | 3 | 2 | 2 | 11
Lymphoedema (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 1
Pallor (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 1
Peripheral artery aneurysm (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 1
Peripheral artery occlusion (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 1
Peripheral artery thrombosis (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 1
Phlebitis (Vascular disorders) | 0 | 1 | 1 | 0 | 1 | 3
Phlebitis superficial (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 1
Poor venous access (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 1
Shock (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of pooled data (i.e.,data from all sites) in clinical trial or disclosure of trial results in their entirety.

DOCUMENTS (2):
  • Statistical Analysis Plan (2014-10-29): https://cdn.clinicaltrials.gov/large-docs/47/NCT00946647/SAP_000.pdf
  • Study Protocol (2016-11-18): https://cdn.clinicaltrials.gov/large-docs/47/NCT00946647/Prot_001.pdf